CLINICAL TRIAL: NCT03969862
Title: Validation Study of Noveos® System as a Diagnostic Tools for Allergy
Brief Title: Validation Study of NOVEOS® System (HYCOR)
Acronym: HYCOR
Status: Terminated | Type: Observational
Why Stopped: Covid-19 sanitary crisis
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hycor Biomedical (Industry)
Responsible Party: Sponsor
Other Study IDs: 7572
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Allergen-mediated IgE Allergy
Keywords: Allergy diagnostic tool; Specific IgE assays; Allergens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with an allergen-mediated IgE allergy: Patients with a clinical history consistent with an allergen-mediated IgE allergy & with a sensitization demonstrated by a positive Prick-Test for the allergen source tested
  Interventions: Device: NOVEOS® system
- Patient without an allergen-mediated IgE allergy: Patient without a clinical history compatible with an IgE allergy-mediated allergy and without PT sensitization to be allergen
  Interventions: Device: NOVEOS® system

INTERVENTIONS:
Device: NOVEOS® system — The NOVEOS® System is a fully automated, high-throughput immunoassay platform that uses magnetic microbeads as a solid phase.
  This is a partially closed system that is primarily intended for the determination of specific IgE with NOVEOS® Hycor allergens. It has the CE mark.

SUMMARY:
Background : The NOVEOS® method is a chemiluminescent immunoassay used to provide quantitative detection of total IgE and allergen-specific IgE antibodies in human serum.

The IgE antibody assay has an essential place in the diagnosis of mediated IgE allergies.

This system could become an alternative to the techniques used today. NOVEOS® uses a quick and convenient method to give results concerning the patient's sensitization profile towards allergens. The volume required for the assays is 4 μl (against more than 100 μl for current techniques), which is particularly important in pediatric and geriatric populations where it may be more difficult to take larger samples.

NOVEOS® also brings true autonomy. In fact, the incorporated reagents provide sufficient capacity for 8 hours of continuous testing.

Objective: Validate the NOVEOS® system as an allergy diagnostic tool, by estimating the sensitivity and specificity of the NOVEOS® assays compared to the gold standard diagnostic represented by the clinical history and PT positive, for a panel of 20 allergens

Methods: This is a validation study of a new immunoassay method (Système NOVEOS®).

The study includes :

* A preliminary phase to familiarize the team with the use of the NOVEOS® system. It is planned to analyze its technical characteristics: the precision, the sensitivity. Eight allergens will be tested, on a cohort of 136 patients
* A validation study of the technique as a diagnostic tool for allergy (sensitivity and specificity compared to the gold standard represented by clinical history and positive PT) and comparison between the new technique and the ImmunoCap® system. Twenty allergens will be tested prospectively, each on 50 cases and 10 controls. A single patient may be both a case for an allergen and a witness for another. For rare allergies, the blood database of the Allergy Service will be used, and affected patients will be contacted to request their non-opposition.

ELIGIBILITY:
IncInclusion criteria:

* Patient who is at least 6 years old
* The patient must be an affiliate or beneficiary of a health insurance plan

Exclusion criteria:

* Patient refusing to take part in the study
* Patient participated in another study that may influence test results
* The patient is in an exclusion period determined by a previous study
* The patient is under the protection of justice, under guardianship or under curatorship
* Patient under antihistaminic H1 treatment preventing the achievement of Prick-tests
* The patient is pregnant
* The patient is breastfeeding
* The patient has a history of tumor, autoimmune, or immune deficiency pathology
* The patient suffers from a hematological pathology (coagulation disorders, anemia) that could interfere with the blood test

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient consulting in our allergy unit for a suspicion of allergy (respiratory, food, drug, hymenoptera venoms)
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the NOVEOS® assay compared to the gold standard diagnosis. | 24 months
  In order to validate the NOVEOS® system as an allergy diagnostic tool, We have to estimate the sensitivity and specificity of the NOVEOS® assays compared to the gold standard diagnostic represented by the clinical history and Prick Test positive, for a panel of 20 allergens.

SECONDARY OUTCOMES:
Specific IgE assessed by NOVEOS® | 24 months
  The serum-specific IgE assay is an in vitro assay of IgE antibodies that are able to bind specifically to their allergen.
  Today, there are techniques that allow the assay of both the IgE reactivity against sources of allergens, but also against the different allergenic components.
  The results of the NOVEOS® method will be considered acceptable according to the following criteria:
  * Total agreement ratio of sample recovery ≥ 0.8
  * Linear Regression / Correlation between the 2 techniques, R ≥ 0.8
Specific IgE assessed by Thermo-Fisher ImmunoCAP® | 24 months
  The serum-specific IgE assay is an in vitro assay of IgE antibodies that are able to bind specifically to their allergen.
  Today, there are techniques that allow the assay of both the IgE reactivity against sources of allergens, but also against the different allergenic components. There are already commercially available, validated and standardized methods; the most used is the Thermo-Fisher ImmunoCAP® (capable of detecting specific IgE amounts> 0.1 kUA / L).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, MD,PHD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No